CLINICAL TRIAL: NCT07082257
Title: Precision Performance Status Compared With ECOG Performance Status- A Pilot Cross Sectional Observational Study
Brief Title: Precision Performance Status Compared With ECOG Performance Status
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-22-6; NCI-2022-09079 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-22-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-07-10; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational ("Get Up and Go" and chair-to-table assessments): Patients undergo "Get Up and Go" assessment as well as a chair-to-table assessment during the clinic visit on study.
  Interventions: Other: Functional Assessment; Behavioral: Timed Get Up and Go Test

INTERVENTIONS:
Other: Functional Assessment — Undergo chair-to-table assessment
Behavioral: Timed Get Up and Go Test — Undergo "Get Up and Go" assessment

SUMMARY:
This study compares consumer movement trackers to the Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) in monitoring cancer patient movement. The ECOG PS emphasizes a patient's ambulatory status (ability to walk around), and scores patients on a scale of 0-5: 0 (no restrictions), 1 (ambulatory), 2 (< 50% of hours spent in bed, unable to carry out work activities), 3 (> 50% of hours spent in bed, limited in self care), 4 (bedbound and gravely disabled) and 5 (deceased). Accurate assessment of a patient's PS is paramount in informing therapeutic decision-making, whether it be to predict response and tolerability to treatment or determine eligibility for clinical trials. However, the ECOG PS scale is observational, and therefore limited in its precision. Information gained in this study may help researchers learn if there is a better way to assess patient movement with computerized analysis tools using movement trackers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the correlation between patient acceleration of the spine base/non-pivoting leg captured with in-office movement trackers, and physician/patient assessed Eastern Cooperative Oncology Group (ECOG) performance status (PS) using a Microsoft Kinect movement tracker.

SECONDARY OBJECTIVES:

I. To determine the correlation between clinician/patient assessed ECOG PS and Kinect assessed ECOG PS score.

II. To determine the range of measured patient acceleration measurements for each ECOG score between 0 and 3.

OUTLINE: This is an observational study.

Patients undergo "Get Up and Go" assessment as well as a chair-to-table assessment during the clinic visit on study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer
* Age >= 18 years
* Ability to understand and the willingness to sign a written informed consent
* Able to ambulate without an assistive device

Exclusion Criteria:

* Missing lower limbs
* Known movement disorder such as Parkinson's disease, choreoathetoid movement disorders, essential tremor if that movement disorder is of sufficient severity to require drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with appointments at University of Southern California (USC)/Norris Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Median acceleration at the Spine Base and non-pivoting leg | Day 1
  The Kinect device will record the participant performing the chair to examination table activity and the Get up and Go activity. This recording will quantify spine and non-pivoting leg mean acceleration during movement onto an examination table and the Get up and Go time. These values will be assessed for a linear or monotonic relationship with Eastern Cooperative Oncology Group (ECOG) scores. If a linear relationship is exhibited the primary objective will be evaluated via a Pearson correlation coefficient. However, the supposition is the data will more likely reflect a monotonic relationship. In this event the primary objective will be evaluated via a Kendall Rank Tau-b correlation coefficient.

SECONDARY OUTCOMES:
Video recording assessed ECOG Performance Status (PS) measurement | Baseline
  The relationship between ECOG PS determined subjectively in clinic and ECOG PS determined by reviewing the Kinect recording will be assessed for a linear or monotonic relationship. However, the supposition is a linear relationship is more likely. A Pearson or Kendall Rank correlation will be utilized accordingly to evaluate a correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Nieva, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California